CLINICAL TRIAL: NCT05135520
Title: A Prospective Randomized Controlled Study of Transvaginal Versus Transabdominal Extraction of Laparoscopically-excised Kidney Specimen (STTELS)
Brief Title: Transvaginal Versus Transabdominal Extraction of Laparoscopically-excised Kidney Specimen
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SNUBH B-2105-687-003
Record Dates: First submitted 2021-11-04; First posted 2021-11-26 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Urologic Neoplasms
Keywords: natural orifice specimen extraction; laparoscopic surgery; transvaginal; female
MeSH Terms: conditions — Urologic Neoplasms

STUDY DESIGN:
Intervention Model Description: Transvaginal specimen extraction vs Transabdominal specimen extraction
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transabdominal specimen extraction (Active Comparator): The outcomes of transabdominal specimen extraction in a classic way in patients who underwent multiport laparoscopic surgery for resection of kidney
  Interventions: Procedure: Transabdominal specimen extraction
- Transvaginal natural orifice specimen extraction (NOSE) (Experimental): The outcomes of transvaginal natural orifice specimen extraction (NOSE) in patients who underwent multiport laparoscopic surgery for resection of kidney
  Interventions: Procedure: Transvaginal natural orifice specimen extraction (NOSE)

INTERVENTIONS:
Procedure: Transvaginal natural orifice specimen extraction (NOSE) — Under general anesthesia, patients who are planned to perform multiport laparoscopic surgery for resection of solid organs including kidney or bladder will undergo Transvaginal NOSE
  Arms: Transvaginal natural orifice specimen extraction (NOSE)
Procedure: Transabdominal specimen extraction — Under general anesthesia, patients who are planned to perform multiport laparoscopic surgery for resection of solid organs including kidney or bladder will undergo transabdominal specimen extraction with incision elongation
  Arms: Transabdominal specimen extraction

SUMMARY:
The aim of this study is to evaluate the outcomes of transvaginal natural orifice specimen extraction (NOSE) in patients who are planning multiport laparoscopic surgery for resection of kidney.

DETAILED DESCRIPTION:
Study design:

This is a prospective, randomized, single center trial. This clinical trial was approved by the Institutional Review Boards.

Study process:

All patients gave informed written consent after being informed of the details of the study. Subjects were randomized into either the experimental group (specimen removal through posterior vagina fornix incision) or control groups (specimen removal through extended abdominal incision). All participants underwent demographic and history taking, laboratory tests, a gynecologic examination to determine whether specimen removal through vagina is possible.

To evaluate cosmesis, patient satisfaction and quality of life VAS (Visual Analogue Scale), SF-12 (Short Form-12) health survey, BIQ (Body Image Questionnaire) and POSAS (the Patient and Observer Scar Assessment Scale) will be sent to the patients 6 months after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are accessible with vaginal approach
* Patients scheduled for laparoscopic resection of kidney for benign or malignant diseases
* Patients with normal cervical cancer screening tests within the last 3 years except inflammatory findings

Exclusion Criteria:

* Patients without sexual intercourse
* Patients who are considered unable to remove specimen through vagina due to narrow introitus in gynecological examination
* Patients who are expected to have severe adhesion due to deep infiltrative endometriosis or previous pelvic surgery history
* Patients with abnormal cervical cancer screening tests
* Patients scheduled to perform concomitant hysterectomy

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2021-11-29 (Estimated); Primary Completion 2022-11-29 (Estimated); Study Completion 2023-11-29 (Estimated)

PRIMARY OUTCOMES:
Patient and Observer Scar Assessment Scale (POSAS) | post-op 1 week
  Cosmetic outcomes of scar assessed by Patient and Observer Scar Assessment Scale (POSAS) 1 week and 8 weeks after surgery. The POSAS is the international validated scar assessment questionnaire that measures quality of the scar from the perspective of both patient and observer.
  observer scar assessment scale (OSAS): good (1) - bad (10)
  - vascularization/ pigmentation/ thickness/ relief/ pliability
  patient scar assessment scale (PSAS): No (1) - Yes (10)
  * Is the scar painful?
  * Is the scar itching?
  * Is the scar color different from the color of your normal skin?
  * Is the stiffness of the scar different from the color of your normal skin?
  * Is the thickness of the scar different from the color of your normal skin?
  * Is the scar more irregular than your normal skin?
Patient and Observer Scar Assessment Scale (POSAS) | post-op 8 weeks
  Cosmetic outcomes of scar assessed by Patient and Observer Scar Assessment Scale (POSAS) 1 week and 8 weeks after surgery. The POSAS is the international validated scar assessment questionnaire that measures quality of the scar from the perspective of both patient and observer.
  observer scar assessment scale (OSAS): good (1) - bad (10)
  - vascularization/ pigmentation/ thickness/ relief/ pliability
  patient scar assessment scale (PSAS): No (1) - Yes (10)
  * Is the scar painful?
  * Is the scar itching?
  * Is the scar color different from the color of your normal skin?
  * Is the stiffness of the scar different from the color of your normal skin?
  * Is the thickness of the scar different from the color of your normal skin?
  * Is the scar more irregular than your normal skin?

SECONDARY OUTCOMES:
Vaginal wound assessment | post-op 1 week
  assessment scale: No (0) - Yes (3) Vaginal bleeding Vaginal discharge Vaginal wound pain
Vaginal wound assessment | post-op 8 weeks
  assessment scale: No (0) - Yes (3) Vaginal bleeding Vaginal discharge Vaginal wound pain
Post-op pain assessment | post-op 2hrs
  Pain assessment with Visual analogue scale: No pain (0) - Worst pain (10)
Post-op pain assessment | post-op 6hrs
  Pain assessment with Visual analogue scale: No pain (0) - Worst pain (10)
Post-op pain assessment | post-op 24hrs
  Pain assessment with Visual analogue scale: No pain (0) - Worst pain (10)
Post-op pain assessment | post-op 48hrs
  Pain assessment with Visual analogue scale: No pain (0) - Worst pain (10)
Female Sexual Function Index (FSFI) questionnaire | post-op 5 months
  Assessment Domain: Desire/ Arousal/ Lubrication/ Orgasm/ Satisfaction/ Pain Full scale score range: min 2.0 - max 36

DOCUMENTS (1):
  • Informed Consent Form (2021-11-20): https://cdn.clinicaltrials.gov/large-docs/20/NCT05135520/ICF_000.pdf